CLINICAL TRIAL: NCT07062744
Title: The Role of Swan-Ganz Catheter in Hemodynamic Resuscitation for Patients With Cardiogenic Shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bach Mai Hospital (Other)
Collaborators: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Thang Pham, Primary investigation, Bach Mai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2025-06-20; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Cardiogenic Shock; Pulmonary Artery Catheter Waveform Interpretation; Hemodynamic Management; Hemodynamic Optimization; Hemodynamic Monitoring; Acute Myocardial Infarction (AMI); Critical Care, Intensive Care; Emergency; Cardio Vascular Disease
Keywords: Swan-Ganz; Pulmonary Artery Catheter; Cardiogenic shock; Hemodynamic management; Invasive hemodynamic; Right Heart Catheter
MeSH Terms: conditions — Shock, Cardiogenic; Emergencies | interventions — Catheterization, Swan-Ganz

STUDY DESIGN:
Intervention Model Description: This is a single-arm clinical trial conducted in an intensive care setting. All enrolled patients diagnosed with cardiogenic shock secondary to acute myocardial infarction will undergo goal-directed hemodynamic resuscitation guided by pulmonary artery catheter (Swan-Ganz) monitoring. The study employs a within-subject design, in which each participant serves as their own temporal control through serial hemodynamic assessments and treatment adjustments. There is no comparator or control group. The protocol includes standardized targets for preload, afterload, cardiac output, and oxygen delivery parameters, with data collected at predefined time points to evaluate hemodynamic response, organ perfusion, and short-term clinical outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Swan-Ganz-Guided Hemodynamic Resuscitation (Experimental): Participants in this arm will undergo invasive hemodynamic monitoring using a Swan-Ganz catheter upon admission to the intensive care unit. Hemodynamic variables, including right atrial pressure (RAP), pulmonary artery pressure (PAP), pulmonary capillary wedge pressure (PCWP), cardiac output (CO), cardiac power output (CPO), and mixed venous oxygen saturation (SvO₂) will be continuously measured and used to guide resuscitation. Management will follow a goal-directed algorithm targeting predefined thresholds for preload, afterload, contractility, and oxygen delivery. All patients will receive standard care for acute myocardial infarction, and no control or comparator arm is included in this study.
  Interventions: Device: Swan-Ganz IQ Pulmonary Arterial catheter; Device: Swan-Ganz IQ catheter

INTERVENTIONS:
Device: Swan-Ganz IQ Pulmonary Arterial catheter — A pulmonary artery catheter (Swan-Ganz catheter) will be inserted via the right internal jugular or subclavian vein using a sterile technique and ultrasound guidance. The catheter is advanced into the pulmonary artery with real-time pressure waveform monitoring to confirm accurate positioning.
  Once inserted, the catheter provides continuous invasive hemodynamic monitoring, including measurements of: Right atrial pressure (RAP), Pulmonary artery pressure (PAP), Pulmonary capillary wedge pressure (PCWP), Cardiac output (CO) by thermodilution, Mixed venous oxygen saturation (SvO₂).
  These parameters are recorded at predefined intervals and used to guide goal-directed hemodynamic resuscitation. Clinical interventions such as vasopressor/inotrope titration, fluid resuscitation, or ventilatory support will be adjusted accordingly. All procedures will follow institutional protocols and safety standards. Complications (e.g., arrhythmias, infection) will be monitored and managed per protocol.
  Other Names: Flow-Directed Cathete; Plumonary Artery Catheter Swan-Ganz; Swan-Ganz catheterization; PAC; Invasive hemodynamic monitoring
Device: Swan-Ganz IQ catheter — A pulmonary artery catheter (Swan-Ganz catheter) will be inserted via the right internal jugular or subclavian vein using a sterile technique and ultrasound guidance. The catheter is advanced into the pulmonary artery with real-time pressure waveform monitoring to confirm accurate positioning.
  Once inserted, the catheter provides continuous invasive hemodynamic monitoring, including measurements of: Right atrial pressure (RAP), Pulmonary artery pressure (PAP), Pulmonary capillary wedge pressure (PCWP), Cardiac output (CO) by thermodilution, Mixed venous oxygen saturation (SvO₂). These parameters are recorded at predefined intervals and used to guide goal-directed hemodynamic resuscitation. Clinical interventions such as vasopressor/inotrope titration, fluid resuscitation, or ventilatory support will be adjusted accordingly. All procedures will follow institutional protocols and safety standards. Complications (e.g., arrhythmias, infection) will be monitored and managed per protocol.
  Other Names: Cardiovascular Diagnostic Catheters; Pulmonary Artery Catheter; Swan-Ganz catheterization; Invasive hemodynamic monitoring

SUMMARY:
This clinical trial examines whether the use of the Swan-Ganz catheter, a specialized pulmonary artery catheter, can improve hemodynamic management and treatment outcomes in patients experiencing cardiogenic shock due to acute myocardial infarction (AMI).

Cardiogenic shock is a critical condition marked by the heart's inability to supply adequate blood to the organs, often resulting from a severe heart attack. Despite advancements in care, the condition remains associated with high mortality. Effective monitoring of cardiovascular status is crucial in guiding timely and tailored treatment decisions.

Participants in this study will undergo advanced hemodynamic monitoring using the Swan-Ganz catheter, which provides continuous data on cardiac output and other key parameters. This information enables physicians to better assess circulatory function and adjust therapies accordingly.

The research will evaluate clinical characteristics, response to treatment, and 30-day outcomes in patients managed with this technique. The study also aims to identify factors associated with successful hemodynamic stabilization and potential complications related to catheter use.

A total of 108 adult patients meeting specific eligibility criteria will be enrolled at Bach Mai Hospital over 3 years. Participation is voluntary, and all patients will continue to receive standard-of-care treatment. All personal and medical data will be handled with strict confidentiality.

DETAILED DESCRIPTION:
This is a clinical trial without a control group; a single-center study evaluates goal-directed hemodynamic optimization using pulmonary artery catheterization (Swan-Ganz catheter) in adult patients with cardiogenic shock secondary to acute myocardial infarction (AMI). Cardiogenic shock is characterized by a sustained systolic blood pressure < 90 mmHg, evidence of end-organ hypoperfusion, and a low cardiac index (< 2.2 L/min/m²) despite adequate filling pressures. In AMI patients, persistent low cardiac output and elevated systemic vascular resistance exacerbate tissue hypoxia, leading to multi-organ dysfunction.

Upon ICU admission, a pulmonary artery catheter will be inserted via the internal jugular or subclavian vein. Continuous measurements of right atrial pressure (RAP), right ventricular pressure, pulmonary artery pressure (PAP), pulmonary capillary wedge pressure (PCWP), cardiac output (via thermodilution), and mixed venous oxygen saturation (SvO₂) will be recorded at baseline and predefined intervals (0, 3, 6, 9, 12, 24 hours). Data will guide titration of inotropes (e.g., dobutamine targeting cardiac index ≥ 2.2 L/min/m²), vasopressors (e.g., norepinephrine to maintain MAP ≥ 65 mmHg), and fluid management (to achieve PCWP from 12 to 18 mmHg and CVP between 8 to 12 mmHg), SvO₂ keep above 60% to 80%, lactat < 2 mmol/L.

The primary endpoint is 30-day all-cause mortality and in-hospital mortality. Secondary endpoints include duration of vasopressor/inotrope support, ICU length of stay, incidence of acute kidney injury, and catheter-related adverse events. Hemodynamic variables will be analyzed for outcomes using multivariate regression to identify predictors of successful hemodynamic stabilization.

All enrolled patients (n ≈ 108) will receive standard AMI care, including early revascularization and guideline-directed medical therapy in conjunction with the study protocol. Data collection, storage, and analysis will comply with Good Clinical Practice and the institution's ethics board requirements. Participation is voluntary, and patients may withdraw at any time without affecting their clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Provided written informed consent to participate in the study.
* Diagnosed with cardiogenic shock due to acute myocardial infarction according to IABP-SHOCK II (2012) criteria:

  * Systolic blood pressure (SBP) < 90 mmHg for at least 30 minutes, or requiring vasopressor agents to maintain SBP > 90 mmHg.
  * Evidence of end-organ hypoperfusion, indicated by at least one of the following: Altered mental status, Urine output < 30 mL/hour, Cold extremities with mottled skin, Serum lactate level > 2 mmol/L.

Exclusion Criteria:

* Presence of cervical cellulitis.
* Inability to identify neck anatomy or history of cervical radiotherapy.
* Coagulopathy (INR > 1.5 and/or platelet count < 50 G/L).
* End-stage chronic diseases, including: Advanced malignancy, advanced-stage HIV, bedridden patients for more than 3 months, decompensated liver cirrhosis (Child-Pugh class C).
* Patients with cardiac arrest or mechanical complications such as myocardial rupture prior to Swan-Ganz catheterization.
* Congenital heart defects or intracardiac shunts. Refusal of participation by the patient or their legal representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality at 30 Days | From the date of Swan-Ganz catheter insertion until the date of death from any cause, assessed up to 30 days
  The proportion of participants who die from any cause within 30 days of Swan-Ganz catheter insertion. Mortality will be determined by review of hospital medical records, ICU documentation, or death certificates.
In-Hospital Mortality | From the date of Swan-Ganz catheter insertion until the hospital discharge date or the in-hospital death date, whichever comes first.
  Proportion of enrolled patients who die from any cause during the index hospitalization after Swan-Ganz catheter insertion. Mortality will be determined by review of hospital medical records, ICU documentation.
Hemodynamic stabilization was achieved within 24 hours | Up to 24 hours after Swan-Ganz catheter insertion
  Proportion of patients achieving predefined hemodynamic targets within 24 hours following Swan-Ganz catheter insertion. Targets include mean arterial pressure (MAP) ≥ 65 mmHg, cardiac index (CI) ≥ 2.2 L/min/m², central venous oxygen saturation (SvO₂) ≥ 60%, pulmonary capillary wedge pressure (PCWP) between 12 and 18 mmHg, and central venous pressure (CVP) between 8 and 12 mmHg.

SECONDARY OUTCOMES:
Length of ICU stay | From the date of ICU admission until the date of ICU discharge, assessed up to 30 days.
  Total number of days from emergency department ICU admission to emergency department ICU discharge for each participant.
Incidence of Catheter-Related Complications | From the date of Swan-Ganz catheter insertion until the date of catheter removal, assessed up to 30 days.
  The incidence of specific complications related to Swan-Ganz catheterization will be assessed, including ventricular arrhythmias, catheter malposition, CLABSI, bleeding at the insertion site, pneumothorax, hematoma, pericardial effusion, pulmonary artery catheter obstruction, thrombosis, and local site complications. Each complication will be reported individually as a percentage of the total study population.
Duration of Mechanical Ventilation (Ventilator Days) | From the date of endotracheal intubation and mechanical ventilation until the date of weaning mechanical ventilation success or death, assessed up to 30 days.
  Number of calendar days that the patient remains on invasive mechanical ventilation from the time of endotracheal intubation until successful extubation or death. Reintubation within 48 hours will be considered part of the same ventilation episode.
Continuous Requirement for Renal Replacement Therapy (CRRT) | From the date of emergency department admission until the date of hospital discharge or death, assessed up to 30 days.
  Proportion of participants who require any form of renal replacement therapy (intermittent hemodialysis, continuous renal replacement therapy, or sustained low-efficiency dialysis) during the index hospitalization for cardiogenic shock.

CONTACTS AND LOCATIONS:
Overall Officials: Thang Xuan Pham, MD, PhD Candidate, Principal Investigator — Hanoi Medical University
Locations (1):
- BachMai Hospital, Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tehrani BN, Truesdell AG, Psotka MA, Rosner C, Singh R, Sinha SS, Damluji AA, Batchelor WB. A Standardized and Comprehensive Approach to the Management of Cardiogenic Shock. JACC Heart Fail. 2020 Nov;8(11):879-891. doi: 10.1016/j.jchf.2020.09.005. PMID 33121700
- [Background] Bertaina M, Galluzzo A, Rossello X, Sbarra P, Petitti E, Prever SB, Boccuzzi G, D'Ascenzo F, Frea S, Pidello S, Morici N, Sacco A, Oliva F, Valente S, De Ferrari GM, Ugo F, Rametta F, Attisani M, Zanini P, Noussan P, Iannaccone M. Prognostic implications of pulmonary artery catheter monitoring in patients with cardiogenic shock: A systematic review and meta-analysis of observational studies. J Crit Care. 2022 Jun;69:154024. doi: 10.1016/j.jcrc.2022.154024. Epub 2022 Mar 25. PMID 35344825
- [Background] Tehrani BN, Truesdell AG, Sherwood MW, Desai S, Tran HA, Epps KC, Singh R, Psotka M, Shah P, Cooper LB, Rosner C, Raja A, Barnett SD, Saulino P, deFilippi CR, Gurbel PA, Murphy CE, O'Connor CM. Standardized Team-Based Care for Cardiogenic Shock. J Am Coll Cardiol. 2019 Apr 9;73(13):1659-1669. doi: 10.1016/j.jacc.2018.12.084. PMID 30947919
- [Background] Chetana Shanmukhappa S, Lokeshwaran S. Venous Oxygen Saturation. 2024 Sep 10. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK564395/ PMID 33232065
- [Background] Kadosh BS, Berg DD, Bohula EA, Park JG, Baird-Zars VM, Alviar C, Alzate J, Barnett CF, Barsness GW, Burke J, Chaudhry SP, Daniels LB, DeFilippis A, Delicce A, Fordyce CB, Ghafghazi S, Gidwani U, Goldfarb M, Katz JN, Keeley EC, Kenigsberg B, Kontos MC, Lawler PR, Leibner E, Menon V, Metkus TS, Miller PE, O'Brien CG, Papolos AI, Prasad R, Shah KS, Sinha SS, Snell RJ, So D, Solomon MA, Ternus BW, Teuteberg JJ, Toole J, van Diepen S, Morrow DA, Roswell RO. Pulmonary Artery Catheter Use and Mortality in the Cardiac Intensive Care Unit. JACC Heart Fail. 2023 Aug;11(8 Pt 1):903-914. doi: 10.1016/j.jchf.2023.04.007. Epub 2023 Jun 14. PMID 37318422
- [Background] Hunziker L, Radovanovic D, Jeger R, Pedrazzini G, Cuculi F, Urban P, Erne P, Rickli H, Pilgrim T; AMIS Plus Registry Investigators are listed in alphabetic order with the names of the local principal investigators. Twenty-Year Trends in the Incidence and Outcome of Cardiogenic Shock in AMIS Plus Registry. Circ Cardiovasc Interv. 2019 Apr;12(4):e007293. doi: 10.1161/CIRCINTERVENTIONS.118.007293. PMID 30943781
- [Background] Kolte D, Khera S, Aronow WS, Mujib M, Palaniswamy C, Sule S, Jain D, Gotsis W, Ahmed A, Frishman WH, Fonarow GC. Trends in incidence, management, and outcomes of cardiogenic shock complicating ST-elevation myocardial infarction in the United States. J Am Heart Assoc. 2014 Jan 13;3(1):e000590. doi: 10.1161/JAHA.113.000590. PMID 24419737
- [Background] Goldberg RJ, Spencer FA, Gore JM, Lessard D, Yarzebski J. Thirty-year trends (1975 to 2005) in the magnitude of, management of, and hospital death rates associated with cardiogenic shock in patients with acute myocardial infarction: a population-based perspective. Circulation. 2009 Mar 10;119(9):1211-9. doi: 10.1161/CIRCULATIONAHA.108.814947. Epub 2009 Feb 23. PMID 19237658
- [Background] Chow JY, Vadakken ME, Whitlock RP, Koziarz A, Ainsworth C, Amin F, McIntyre WF, Demers C, Belley-Cote EP. Pulmonary artery catheterization in patients with cardiogenic shock: a systematic review and meta-analysis. Can J Anaesth. 2021 Nov;68(11):1611-1629. doi: 10.1007/s12630-021-02083-2. Epub 2021 Aug 17. PMID 34405356
- [Background] Rea ABBAC, Mihajlovic V, Vishram-Nielsen JKK, Brahmbhatt DH, Scolari FL, Wang VN, Nisar M, Fung NL, Otsuki M, Billia F, Overgaard CB, Luk A. Pulmonary Artery Catheter Usage and Impact on Mortality in Patients With Cardiogenic Shock: Results From a Canadian Single-Centre Registry. Can J Cardiol. 2024 Apr;40(4):664-673. doi: 10.1016/j.cjca.2023.12.005. Epub 2023 Dec 12. PMID 38092192
- [Background] Bertaina M, Galluzzo A, Morici N, Sacco A, Oliva F, Valente S, D'Ascenzo F, Frea S, Sbarra P, Petitti E, Prever SB, Boccuzzi G, Zanini P, Attisani M, Rametta F, De Ferrari GM, Noussan P, Iannaccone M. Pulmonary Artery Catheter Monitoring in Patients with Cardiogenic Shock: Time for a Reappraisal? Card Fail Rev. 2022 Apr 26;8:e15. doi: 10.15420/cfr.2021.32. eCollection 2022 Jan. PMID 35541286
- [Background] Thiele H, Zeymer U, Thelemann N, Neumann FJ, Hausleiter J, Abdel-Wahab M, Meyer-Saraei R, Fuernau G, Eitel I, Hambrecht R, Bohm M, Werdan K, Felix SB, Hennersdorf M, Schneider S, Ouarrak T, Desch S, de Waha-Thiele S; IABP-SHOCK II Trial (Intraaortic Balloon Pump in Cardiogenic Shock II) Investigators; IABP-SHOCK II Investigators. Intraaortic Balloon Pump in Cardiogenic Shock Complicating Acute Myocardial Infarction: Long-Term 6-Year Outcome of the Randomized IABP-SHOCK II Trial. Circulation. 2019 Jan 15;139(3):395-403. doi: 10.1161/CIRCULATIONAHA.118.038201. Epub 2018 Nov 11. PMID 30586721
- [Background] van Diepen S, Katz JN, Albert NM, Henry TD, Jacobs AK, Kapur NK, Kilic A, Menon V, Ohman EM, Sweitzer NK, Thiele H, Washam JB, Cohen MG; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Mission: Lifeline. Contemporary Management of Cardiogenic Shock: A Scientific Statement From the American Heart Association. Circulation. 2017 Oct 17;136(16):e232-e268. doi: 10.1161/CIR.0000000000000525. Epub 2017 Sep 18. PMID 28923988
- [Background] Garan AR, Kanwar M, Thayer KL, Whitehead E, Zweck E, Hernandez-Montfort J, Mahr C, Haywood JL, Harwani NM, Wencker D, Sinha SS, Vorovich E, Abraham J, O'Neill W, Burkhoff D, Kapur NK. Complete Hemodynamic Profiling With Pulmonary Artery Catheters in Cardiogenic Shock Is Associated With Lower In-Hospital Mortality. JACC Heart Fail. 2020 Nov;8(11):903-913. doi: 10.1016/j.jchf.2020.08.012. PMID 33121702
- [Background] Yoo TK, Miyashita S, Davoudi F, Imahira U, Al-Obaidi A, Chweich H, Huggins GS, Kimmelstiel C, Kapur NK. Clinical impact of pulmonary artery catheter in patients with cardiogenic shock: A systematic review and meta-analysis. Cardiovasc Revasc Med. 2023 Oct;55:58-65. doi: 10.1016/j.carrev.2023.04.008. Epub 2023 Apr 17. PMID 37100652
- [Background] Sinha SS, Rosner CM, Tehrani BN, Maini A, Truesdell AG, Lee SB, Bagchi P, Cameron J, Damluji AA, Desai M, Desai SS, Epps KC, deFilippi C, Flanagan MC, Genovese L, Moukhachen H, Park JJ, Psotka MA, Raja A, Shah P, Sherwood MW, Singh R, Tang D, Young KD, Welch T, O'Connor CM, Batchelor WB. Cardiogenic Shock From Heart Failure Versus Acute Myocardial Infarction: Clinical Characteristics, Hospital Course, and 1-Year Outcomes. Circ Heart Fail. 2022 Jun;15(6):e009279. doi: 10.1161/CIRCHEARTFAILURE.121.009279. Epub 2022 May 5. PMID 35510546
- [Background] Lim HS. Cardiac Power Output Revisited. Circ Heart Fail. 2020 Oct;13(10):e007393. doi: 10.1161/CIRCHEARTFAILURE.120.007393. Epub 2020 Sep 30. No abstract available. PMID 32993372
- [Background] Fincke R, Hochman JS, Lowe AM, Menon V, Slater JN, Webb JG, LeJemtel TH, Cotter G; SHOCK Investigators. Cardiac power is the strongest hemodynamic correlate of mortality in cardiogenic shock: a report from the SHOCK trial registry. J Am Coll Cardiol. 2004 Jul 21;44(2):340-8. doi: 10.1016/j.jacc.2004.03.060. PMID 15261929

DOCUMENTS (3):
  • Study Protocol (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT07062744/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT07062744/SAP_001.pdf
  • Informed Consent Form (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT07062744/ICF_002.pdf